CLINICAL TRIAL: NCT01642576
Title: Comparing Effects of Diet, With or Without Exercise, on Sexual, Urinary and Endothelial Function, Inflammatory Profile and Quality of Life in Obese Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZCHOENFU
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Sexual Dysfunction; Endothelial Dysfunction; Quality of Life; Inflammation
Keywords: obesity; men; sexual function; urinary tract symptoms; endothelial function; inflammation; quality of life
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Inflammation; Obesity; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- diet modification (Experimental): counselling on caloric restriction and healthy eating
  Interventions: Behavioral: weight loss counselling
- weight management program (Experimental): dietician and sports trainer, physician counselling on weight loss
  Interventions: Behavioral: weight loss counselling

INTERVENTIONS:
Behavioral: weight loss counselling — Diet counselling with or without sports trainers, over 8 months

SUMMARY:
This study aims to compare the effects of 8 months of diet modification, with or without exercise, on weight loss, sexual, urinary and endothelial function, systemic inflammation and quality of life in obese men.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 30-65 years
* Body Mass Index (BMI) >/= 27.5 kg/m2
* Waist circumference (WC) >/= 90 cm

Exclusion Criteria:

* pituitary disease or cranial radiotherapy
* previous or current androgen replacement or deprivation therapy
* current treatment for sexual problems or LUTS
* glomerular filtration rate < 60 ml/min
* liver disease
* alcohol intake exceeding 500 g/week in the previous 12 months
* use of opiates, glucocorticoids, recreational drugs or phosphodiesterase inhibitors

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
erectile function | 8 months
  IIEF-5 score

SECONDARY OUTCOMES:
lower urinary tract symptoms | 8 months
  IPSS score

CONTACTS AND LOCATIONS:
Overall Officials: Joan Khoo, MRCP, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore, Singapore